CLINICAL TRIAL: NCT05422911
Title: A Phase 2 Randomized Study of YONSA® (Abiraterone Acetate), Enzalutamide or Apalutamide as First Line Therapy in Veterans With Castrate-sensitive Prostate Cancer
Brief Title: Abiraterone, Enzalutamide, or Apalutamide in Castrate-sensitive Prostate Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Bates, Oncologist, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1641701
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Cancer; Neoplasm, Prostate
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abiraterone Acetate (Active Comparator)
  Interventions: Drug: Abiraterone acetate
- Standard of Care (Active Comparator)
  Interventions: Drug: Apalutamide; Drug: Enzalutamide

INTERVENTIONS:
Drug: Abiraterone acetate — YONSA® (abiraterone acetate), YONSA® 500 mg (four 125 mg tablets) or 625 mg (five 125 mg tablets) administered orally once daily in combination with methylprednisolone 4 mg administered orally twice daily + physician's choice GnRH agonist/antagonist [unless the Veteran has had prior bilateral orchiectomy].
  Arms: Abiraterone Acetate
Drug: Apalutamide — Apalutamide, 240 mg (four 60 mg tablets) administered orally once daily + physician's choice GnRH agonist/antagonist [unless the Veteran has had prior bilateral orchiectomy].
  Arms: Standard of Care
Drug: Enzalutamide — Enzalutamide, 160 mg (four 40 mg capsules) administered orally once daily + physician's choice GnRH agonist/antagonist [unless the Veteran has had prior bilateral orchiectomy].
  Arms: Standard of Care

SUMMARY:
The investigators have used national VHA data to demonstrate real-world efficacy of abiraterone and enzalutamide in Veterans with mCRPC. In the real-world that is the VHA, the investigators have successfully estimated g values that accurately predict OS and the use of this metric in other settings should now be explored. In the egalitarian system that is the VHA the treatment of prostate cancer is excellent, uniform across the US and indifferent to race. The choices made are clearly personalized, given not all men received all therapies and that younger Veterans were treated more aggressively.

But with survivals that rival those in registration trials that enroll optimally fit individuals usually not encumbered by the co-morbidities that afflict many Veterans, the outcomes are testimony to the fact that for this common malady of older Veterans with whom VA physicians have broad experience the care administered is unsurpassed. Importantly this care at least as regards Veterans with mCRPC demonstrates that given equal access to health care, African Americans with prostate cancer fared as well if not better than Caucasians and importantly had better outcomes with abiraterone, an observation needing further exploration as these therapies move up front.

ELIGIBILITY:
Inclusion Criteria:

* Veterans must meet the following to be eligible to participate:
* Be willing and able to provide written informed consent for the trial.
* Age ≥18 years of age on day of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (on a scale from 0 to 5, with higher scores indicating greater disability and a score of 5 indicating death).
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, signet-cell features, or small-cell features in either a recently obtained sample or in the archival sample at the time of diagnosis.
* Have been receiving or will receive androgen-deprivation therapy with a gonadotropin releasing hormone agonist or antagonist or have undergone bilateral orchiectomy (i.e., medical, or surgical castration).
* High risk for the development of progression of disease/metastasis, defined as (i) a minimum of three rising PSA values (PSA1 < PSA2 < PSA3) at an interval of at least 1 week apart; (ii) a PSA level of 2 ng per milliliter (2 μg/L) or greater; and (iii) a PSA doubling time of 9 months or less during continuous androgen-deprivation therapy (bilateral orchiectomy or treatment with gonadotropin-releasing hormone analogue agonists or antagonists) as calculated with the use of the method of Pound et al.
* Has not received abiraterone acetate, enzalutamide, or apalutamide at the time of enrollment.
* Have a predicted life expectancy of >12 months.
* For patients receiving bisphosphonates or denosumab, dose must be stable for at least 4 weeks before randomization.
* Able to swallow the study drug and comply with study requirements.
* Laboratory tests meet minimum safety requirements:

  * Hepatic: AST ≤2.5 X institutional ULN, ALT ≤2.5 X institutional ULN
  * Renal: Creatinine clearance ≥30 ml/min or serum creatinine ≤1.8 mg/dl
  * Hematological: Absolute neutrophil count ≥1000/mm3, Platelet count ≥100,000/mm3; Hemoglobin >9 g/dL Note: The presence of metastatic disease as assessed by any modality is not a contraindication for enrollment.

Exclusion Criteria:

Subjects with any of the following will not be enrolled:

* Prior cytotoxic chemotherapy, aminoglutethimide, ketoconazole, abiraterone acetate, apalutamide or enzalutamide for the treatment of prostate cancer or participation in a clinical trial of an investigational agent that inhibits the androgen receptor or androgen synthesis (unless treatment was placebo).
* Treatment with hormonal therapy (e.g., androgen receptor inhibitors, estrogens, 5-alpha reductase inhibitors) or biologic therapy for prostate cancer (other than approved bone targeting agents and GnRH agonist/antagonist therapy) within 4 weeks of randomization
* Other malignancy except: (a) Subjects who have been successfully treated and are disease free for 3 years; (b) a history of completely resected non-melanoma skin cancer; or (c) successfully treated in situ carcinoma.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma).
* Deep vein thrombosis or pulmonary embolism in the past 3 months that in the opinion of the physician makes the patient medically unstable.
* Patients who are receiving any other investigational agents concurrently.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PSA Progression | 2 years
  Primary Objectives
  1. In Veterans with castrate-sensitive prostate cancer demonstrate that administration of YONSA® (abiraterone acetate) first is not inferior to the administration of physician's choice enzalutamide or apalutamide first with efficacy measured by the rate (g) of tumor growth based on PSA measurement.
  2. In Veterans with castrate-sensitive prostate cancer demonstrate that the efficacy of abiraterone acetate is superior in African American compared to Caucasian Veterans with efficacy measured by the rate (g) of tumor growth based on PSA determination.

SECONDARY OUTCOMES:
PSA Response | 2 years
  PSA response based Prostate Cancer Working Group 2 guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No